CLINICAL TRIAL: NCT07064967
Title: Non-Helium Magnetoencephalography for Identifying Neurobiological Features and Functional Biomarkers in Children With Autism Spectrum Disorder: An Observational Cohort Study
Brief Title: Non-Helium Magnetoencephalography in Autism Spectrum Disorder
Status: Recruiting | Type: Observational
Sponsor: Guangzhou Women and Children's Medical Center (Other)
Collaborators: Beijing X-Magtech Technology Limited (Unknown)
Responsible Party: Sponsor
Other Study IDs: 447A01
Record Dates: First submitted 2025-07-03; First posted 2025-07-15 (Actual); Last update posted 2025-07-15 (Actual); Status verified 2024-11

CONDITIONS: Autism Spectrum Disorder (ASD)
Keywords: Autism Spectrum Disorder; Magnetoencephalography
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — Magnetoencephalography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ASD: Participants in the ASD group consisted of children diagnosed with Autism Spectrum Disorder according to DSM-5 criteria.
  Interventions: Diagnostic Test: Magnetoencephalography
- Control: Participants in the Control group consisted of typically developing children.
  Interventions: Diagnostic Test: Magnetoencephalography

INTERVENTIONS:
Diagnostic Test: Magnetoencephalography — Participants will undergo magnetoencephalography scan in both resting and tasking state.

SUMMARY:
The goal of this observational study is to learn how brain activity in children with autism spectrum disorder (ASD) differs from typical developing children using magnetoencephalography (MEG).

The main questions this study aims to answer are:

Do children with ASD show different patterns of neural oscillation compared to typically developing children? Can MEG identify specific brain features that help ASD diagnosis?

Participants will undergo MEG scan in both resting and tasking state, and their brain activity will be analyzed for characteristic neural oscillations and connectivity patterns.

This study may help develop better tools for early ASD diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Boys aged 6 to 12 years;
* Diagnosis of Autism Spectrum Disorder meeting DSM-5 criteria;
* Intelligence quotient (IQ) score > 70 (assessed via Wechsler Intelligence Scale for Children or other validated cognitive test);
* Sufficient compliance to participate in MEG experiments.

Exclusion Criteria:

* Comorbid neurological disorders, genetic syndromes, or severe developmental disabilities;
* Metallic implants that may interfere with MEG signal acquisition;
* Current use of antipsychotic medications or sedatives.

Ages: 6 Years to 12 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Pediatric patients of Guangzhou Women and Children's Medical Center
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Identification of Neural Oscillation Characteristics in Children with Autism Spectrum Disorder | Baseline assessment (single time point, within 1 week of enrollment).
  The primary outcome will measure group differences in neural oscillation features (e.g., spectral power and spatial distribution) across frequency bands (alpha, beta, gamma) between children with Autism Spectrum Disorder and typically developing children during resting-state and task-based conditions. Quantified using time-frequency analysis of magnetoencephalography data. Statistical analysis will include independent t-tests (or Mann-Whitney U tests for non-normally distributed data) with false discovery rate (FDR) correction, using SPSS version 27.0.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Women and Children's medical center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No